CLINICAL TRIAL: NCT06991543
Title: Structural Heat Adaptation and Education in Urban Setting (SHAPES Trial)
Brief Title: Structural Heat Adaptation and Education in Urban Setting
Acronym: SHAPES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University College, London (Other)
Responsible Party: Principal Investigator, Dr Jai Kumar Das, Associate Professor, Associate Director, Institute for Global Health and Development, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11548; 226752/Z/22/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2025-05-06; First posted 2025-05-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Heat Illness; Quality of Life
Keywords: heat illness; behaviour modification; personal cooling; Structural modification; heat adaptation; prevention; quality of life
MeSH Terms: conditions — Heat Stress Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience and Heat Adaptation Bundle (Experimental): Intervention Arm: Resilience and Heat Adaptation Bundle (ReHAB):
  The ReHAB consists of three components; community education and awareness, personal lifestyle and cooling behavior modification, and participatory local structural and environmental heat mitigation solutions. The behavioral and educational interventions will be delivered through community mobilization whereas structural interventions will encompass modifications in the existing structures to lower the indoor ambient temperature and reduce heat effects.
  Interventions: Behavioral: Community education and awareness, and personal lifestyle and cooling behavior modification; Other: Participatory local structural and environmental heat mitigation solutions
- Control (No Intervention): The control arm will not receive any intervention.

INTERVENTIONS:
Behavioral: Community education and awareness, and personal lifestyle and cooling behavior modification — This component of the ReHAB will be achieved through community mobilization, which will encompass awareness and motivational activities throughout the intervention duration. Community groups (CGs) will be formed in each of the 11 clusters. Both male and female CGs will be formed separately and will be responsible for community mobilization activities, surveillance for primary outcome. Each CG will comprise of 6-8 members and will be a diverse group of people with varying qualifications, including local government members, local elders/elites, religious leaders, and prominent male and female members of the community. they could also name their respective CGs to enhance association, identity, and affiliation. These CGs will facilitate culturally tailored workshops, dissemination of early warnings regarding heat waves, awareness sessions, and door-to-door outreach focused on heat-health fundamentals. CGs will also maintain simple logbooks to track any incidence of heat related illness.
  Other Names: behavioral change; early warning system
  Arms: Resilience and Heat Adaptation Bundle
Other: Participatory local structural and environmental heat mitigation solutions — Participatory local structural and environmental heat mitigation solutions will be delivered through community participatory approach where the community and project will share the cost of intervention to improve ownership. This contribution can be monetary or non-monetary, for example, provision of labor or supplies. The modifications include:
  1. Paints (Solar Reflective Paints, Lime Paints)
  2. Shading (Façade, Roof)
  3. Energy Sufficiency (Solar Panels with complete accessories)
  4. Community Shading (Plantation, Street Shading, Field Shading space)
  5. Ventilation (Windows, Wind catchers)
  Arms: Resilience and Heat Adaptation Bundle

SUMMARY:
This study aims to understand whether simple, low-cost interventions, such as improved home cooling, practical advice, and minor home modifications, can help protect people's health and improve quality of life during periods of extreme heat in densely populated, low-income neighborhoods of Karachi, Pakistan.

Key Questions the Study Seeks to Answer:

1. Can these interventions reduce heat-related health problems such as dizziness, headaches, and heatstroke and improve the quality of life?
2. Can they lower indoor temperatures and improve sleep quality, comfort, and daily functioning?

To answer these questions, researchers will compare communities where families receive heat-related support and information with similar communities that do not, to assess any differences in health and well-being.

What Participants Can Expect:

* Answer questions about their health, living conditions, and how they cope with heat
* Have small temperature sensors placed inside their homes
* Some participants may wear a lightweight wristband that tracks sleep and heart rate
* In selected households, cooling improvements will be made, such as adding shade, applying reflective roof paint, or enhancing airflow

Purpose:

This study seeks to identify affordable and effective strategies to help families stay safe during extreme heat, and to use these insights to support other vulnerable communities facing similar challenges.

ELIGIBILITY:
Inclusion Criteria:

* All households within the selected clusters who provide consent.

Exclusion Criteria:

* Households planning to move away from the study site within the next 6 months
* Individuals with severe mental or physical health conditions that preclude participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7128 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Heat-Related Illness | from baseline to 24 months
  Heat-related illness is defined as any condition resulting from prolonged heat exposure, including heat stroke, heat exhaustion, heat syncope, heat cramps, or heat rash. Data will be collected through weekly household surveillance, and community group reports
Quality of Life Enhancement | 4 month, 7 month, 16 month, 19 month
  Change in the WHOQOL-BREF overall score (mean of domain scores) during two consecutive peak summer and winter seasons

SECONDARY OUTCOMES:
All-cause mortality (Number of Deaths from Any Cause) | from baseline to 24 months
  All-cause mortality refers to the total number of deaths from any cause among trial participants during the study period, confirmed via household visits and healthcare facility records.
Number of Participants with At Least One Hospital Visit During Study Period | During summer months for 2 years
  Defined as the number of participants who visited a secondary or tertiary healthcare facility for any reason during the study period, confirmed by self-report and facility-based records.
Number of Participants Hospitalized for at Least 24 Hours | During summer months for 2 years
  Defined as the number of participants who were admitted to a hospital for at least 24 consecutive hours during the study period, verified through hospital admission records and participant reports.
Change in Self-Reported Thermal Comfort Score | from baseline to 24 months
  Thermal comfort will be assessed using a modified version of the CHEQ-5 thermal comfort survey. Participants rate their satisfaction with indoor thermal conditions. The scale ranges from 1 (very uncomfortable) to 5 (very comfortable). Higher scores indicate better thermal comfort. Assessments will be conducted at baseline, and then monthly afterwards.
Change in Indoor Heat Index | From intervention delivery to 24 months
  Measured as the difference in average indoor heat index before and after intervention using fixed indoor temperature loggers (iButton sensors or Temp-U data loggers). Data collected continuously throughout the study.

OTHER OUTCOMES:
Personalized Heat Exposure (°C) | During summer months for 2 years
  Defined as the average temperature experienced by an individual, measured continuously using wearable temperature monitors. Data will be collected across both indoor and outdoor settings for each participant.
Change in Heart Rate (Beats per Minute) | During summer months for 2 years
  Heart rate will be measured using Fitbit Inspire 3 devices. Data are recorded at hourly intervals. The outcome will be reported as the change in average heart rate from baseline to follow-up.
Sleep quality | During summer months for 2 years
  Sleep quality will be assessed using Fitbit Inspire 3, which detects sleep stages (REM, light, deep) and wakefulness. Data include total sleep time, sleep efficiency, and time spent in each stage. Higher efficiency and longer sleep duration indicate better sleep quality.
Physical Activity Level Based on Daily Step Count and Activity Classification | During summer months for 2 years
  Measured using Fitbit Inspire 3 devices. Participants will be categorized as sedentary, lightly active, moderately active, or very active based on daily movement data (step counts, active minutes). Categories follow Fitbit's proprietary activity classification algorithm.
Total Daily Energy Expenditure (Kilocalories) | During summer months for 2 years
  Measured using Fitbit Inspire 3. This includes calories burned through basal metabolic rate and physical activity. Reported as the average number of kilocalories burned per day per participant.

CONTACTS AND LOCATIONS:
Overall Officials: jai K Das, Principal Investigator — Institute for global health and development, Aga Khan University.
Locations (1):
- Bilal Colony, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Upon reasonable request.